CLINICAL TRIAL: NCT02938312
Title: Deep South Network for Cancer Control - Healthier Weight Among African American Women
Brief Title: Journey to Better Health
Acronym: JTBH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Monica L Baskin, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F100708003; 1U54CA153719 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight Loss Only (Active Comparator): 24- month weight loss program (year 1: weekly in-person meetings for 6 months, followed by 2 meetings per month for 3 months, then monthly for 3 months; year 2: monthly phone calls)
  Interventions: Behavioral: Weight Loss Only
- Weight Loss Plus (Experimental): Same intervention as "Weight Loss Only" but includes community-wide interventions to increase access to healthy affordable food and opportunities for safe and convenient physical activity
  Interventions: Behavioral: Weight Loss Plus

INTERVENTIONS:
Behavioral: Weight Loss Only — Participants will attend in-person weekly sessions (about 1.5 hours each) for 6 months and then twice a month for 3 months and monthly for 3 months. Sessions focus on behavioral techniques supporting healthy diet (including calorie restriction for weight loss) and achieving recommended amounts of physical activity per week. During 1-year weight loss maintenance, participants receive monthly motivational phone calls.
  Arms: Weight Loss Only
Behavioral: Weight Loss Plus — Participants attend in-person meetings as described above. This condition also includes community-wide strategies to increase access to healthy affordable food and safe opportunities for physical activity.
  Arms: Weight Loss Plus

SUMMARY:
This study is being conducted in 8 rural counties in Alabama and Mississippi (4 per state). Approximately 400 overweight or obese African American women living in the selected counties will participate in a 2-year weight loss study.

DETAILED DESCRIPTION:
Using a cluster-randomized study design, 400 overweight or obese African American women living in 8 rural counties in Alabama and Mississippi associated with the Deep South Network for Cancer Control will be assigned to either a weight loss only or weight loss plus community strategies condition for 2 years.

Weight Loss Only condition: In year 1, participants will attend weekly in-person group sessions (1.5 hours each) aimed at behavioral changes for weight loss (diet and physical activity) for 6 months followed by twice a month meetings for 3 months, then monthly meetings for 3 months. In year 2, monthly phone calls will be used to encourage continued behavior change or weight maintenance. In-person group meetings will be facilitated by a trained lay staff and community health advisors. Monthly phone calls will be conducted by the community health advisor.

Weight Loss Plus Community Strategies condition: Participants will receive the same weight loss program as the Weight Loss Only condition. In addition, a community-based organization or other non-profit group in the targeted community will receive funds and technical assistance to implement community-wide efforts to increase access to healthy affordable food and safe and convenient opportunities for physical activity (e.g., increase farmer's markets, develop walking trails).

Over the course of the study, participants will complete four full assessments to include measurement of height and weight (to calculate BMI), waist circumference, blood pressure, finger-stick blood draw for lipid and glucose testing, dietary recall, and questionnaires concerning participation in physical activity, self-efficacy for eating and exercise behaviors, depressive symptoms, perceived stress, social support, and demographic information (e.g., age, marital status, education, employment, household income).

ELIGIBILITY:
Inclusion Criteria:

* African American female
* Live or work in target county
* BMI >= 25 kg/m2

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next year
* Known major medical or psychological condition known to influence body weight
* Uncontrolled hypertension (BP > 160 mmHg systolic or >100 mmHg diastolic)
* Cardiovascular event in the preceding 12 months
* History of gastric bypass surgery
* History of psychiatric hospitalization in past 2 years
* History of substance abuse or eating disorder
* Any other condition by which a medical professional has suggested diet modification
* Physical activity and/or weight reduction would be contraindicated

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2010-08; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Weight | baseline to 6-months
  Measured weight (nearest kg)

SECONDARY OUTCOMES:
Waist Circumference | baseline to 6-months
  Measured circumference (nearest cm)
Blood Pressure | baseline to 6-months
  Measured blood pressure (mmHG) - systolic and diastolic
Lipids | baseline to 6-months
  Measured lipids - total cholesterol (mg/dL), Triglycerides (mg/dL), HDL, LDL, ratio
Weight | baseline to 12-months
  Measured weight (nearest kg)
Weight | baseline to 24-months
  Measured weight (nearest kg)
Social Support for Healthy Eating and Exercise | baseline to 6-months
  Self-report questionnaire about perceived level of family and friend support for healthy eating and exercise. Composite and subscale scores are calculated.
Social Support for Healthy Eating and Exercise | baseline to 12-months
  Self-report questionnaire about perceived level of family and friend support for healthy eating and exercise. Composite and subscale scores are calculated.
Social Support Healthy Eating and Exercise | baseline to 24-months
  Self-report questionnaire about perceived level of family and friend support for healthy eating and exercise. Composite and subscale scores are calculated.
Self Efficacy for Healthy Eating and Exercise | baseline to 6-months
  Self-report questionnaire about confidence in ability to eat healthy and exercise. Composite and subscale scores are calculated.
Self Efficacy for Healthy Eating and Exercise | baseline to 12-months
  Self-report
Self Efficacy for Healthy Eating and Exercise | baseline to 24-months
  Self-report questionnaire about confidence in ability to eat healthy and exercise. Composite and subscale scores are calculated.
Dietary Intake | baseline to 6-months
  24 hour recall
Dietary Intake | baseline to 12-months
  24 hour recall
Dietary Intake | baseline to 24-months
  24 hour recall
Perceived Stress Scale | baseline to 6-months
  Self-report questionnaire about frequency of select stressful events. Composite score is calculated based on responses.
Perceived Stress Scale | baseline to 12-months
  Self-report questionnaire about frequency of select stressful events. Composite score is calculated based on responses.
Perceived Stress Scale | baseline to 24-months
  Self-report questionnaire about frequency of select stressful events. Composite score is calculated based on responses.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No